CLINICAL TRIAL: NCT03743389
Title: Application Study of 12G Pigtail Catheter Used for Post-operative Drainage After Thoracoscopic Surgery for Mediastinal Nodes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJTS-CT001
Record Dates: First submitted 2018-09-27; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-09

CONDITIONS: Mediastinal Nodes
Keywords: uniportal video-assisted thoracoscopic surgery; mediastinal nodes; chest drainage; pigtail catheter

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12G pigtail catheter (Experimental)
  Interventions: Device: 12G pigtail catheter
- 16F chest tube (Active Comparator)
  Interventions: Device: 16F chest tube

INTERVENTIONS:
Device: 12G pigtail catheter — 12G pigtail catheter would be used for post-operative chest drainage after uniportal-VATS for mediastinal nodes resection when comparing with the traditional 16F chest tube.
  Arms: 12G pigtail catheter
Device: 16F chest tube — 16F chest tube would be used for post-operative chest drainage after uniportal-VATS for mediastinal nodes resection when comparing with 12G pigtail catheter.
  Arms: 16F chest tube

SUMMARY:
Pigtail catheter(PC) has been used for thoracic drainage in the patients with pneumothorax or traumatic hemothorax/hemopneumothorax, and some study indicated that PC could obtain similar outcomes when comparing with chest tube(CT). Although PC could drain air and fluid out from pleural cavity and also help pulmonary re-expanding, rare reports are available to thoracic post-operative management. Uniportal video-assisted thoracoscopic surgery(VATS) has been widely applied in many medical center in recent years, most of mediastinal nodes could be resected under uniportal-VATS. This study aims to further study the application of 12G PC during post-operative management and comparing the validity and safety between PC(12G) and CT(16F) after uniportal-VATS for mediastinal nodes resection.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 80 years of age.
2. Diagnosed with potentially resectable mediastinal mass.
3. With indication for uniportal-VATS.
4. For whom informed consent will be obtained before the study.

Exclusion Criteria:

1. Previous thoracic surgery at the same side.
2. Have to receive open surgery although uniportal-VATS is planned.
3. Pregnancy.
4. Refuse to sigh the consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
total drainage volume | 1 month
tube duration | 1 month

SECONDARY OUTCOMES:
post-operative pain | 3 days after operation
  assessed via the "Visual Analogue Scale" (VAS) which ranging from 0 (no pain) to 10 (worst imaginable pain).
rate of subcutaneous emphysema | 1 month
infection rate of incision | 1 month
length of hospital stay after surgery | 1 month
rate of chest tube re-insertion or thoracocentesis | 1 month
satisfaction of the incision after healing | 1 month
  Patients would be asked if they are satified with the appearence of the healed incision at the one-month follow-up evalution.